CLINICAL TRIAL: NCT01928524
Title: Phase I Trial With Docetaxel, Oxaliplatin and S1 as First-line Treatment for Patients With Non-resectable Adenocarcinoma of the Esophagus or Gastric
Brief Title: Chemotherapy for Patients With Cancer of the Stomach
Acronym: DOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KFE 12.17
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: First-line Treatment for Patients With Non-resectable Gastric Cancer or Cancer of the Esophagus or
Keywords: Gastric cancer; Cancer of the esophagus; Oxaliplatin; Docetaxel; S1
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Two parallel phase 1/2a studies with 3+3 design with either DOS given every second week or every third week in Caucasian patients (Table 1). Patients were included into DOS2w and DOS3w in sequence.
  In the DOS2w group: Patients received escalating doses of Docetaxel (30-50 mg/m2 on Day 1), fixed doses of O (70 mg/ m2 on Day 1) and S-1 (30-35 mg/m2/day twice daily orally on Days 1-7) every two weeks. In the DOS3w group: Patients received escalating doses of docetaxel (40-60 mg/m2 on Day 1), fixed doses of O (100 mg/ m2 on Day 1) and S-1 (25 mg/m2/day twice daily orally on Days 1-14) every three weeks.
Oversight: Data Monitoring Committee: No

ARMS (7):
- DOS2W Dose level 1A (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2 weeks.
  Interventions: Drug: DOS2w Dose level 1A
- DOS2W Dose level 2A (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2 weeks.
  Interventions: Drug: DOS2w Dose level 2A
- DOS2W Dose level 3A (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2 weeks.
  Interventions: Drug: DOS2w Dose level 3A
- DOS2W Dose level 4A (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2 weeks.
  Interventions: Drug: DOS2w Dose level 4A
- DOS3W Dose level 1B (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3 weeks.
  Interventions: Drug: DOS3w Dose level 1B
- DOS3W Dose level 2B (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3 weeks.
  Interventions: Drug: DOS3w Dose level 2B
- DOS3W Dose level 3B (Experimental): Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3 weeks.
  Interventions: Drug: DOS3w Dose level 3B

INTERVENTIONS:
Drug: DOS2w Dose level 1A — Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (60 mg/2) will be given every 2 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS2w 1A
  Arms: DOS2W Dose level 1A
Drug: DOS2w Dose level 2A — Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS2w 2A
  Arms: DOS2W Dose level 2A
Drug: DOS2w Dose level 3A — Docetaxel (40 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS2w 3A
  Arms: DOS2W Dose level 3A
Drug: DOS2w Dose level 4A — Docetaxel (50 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS2w 4A
  Arms: DOS2W Dose level 4A
Drug: DOS3w Dose level 1B — Docetaxel (40 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS3w 1B
  Arms: DOS3W Dose level 1B
Drug: DOS3w Dose level 2B — Docetaxel (50 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS3w 2B
  Arms: DOS3W Dose level 2B
Drug: DOS3w Dose level 3B — Docetaxel (60 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3 weeks. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
  Other Names: DOS3w 3B
  Arms: DOS3W Dose level 3B

SUMMARY:
The purpose of this study is to determine maximal tolerable dose (MTD) of the combination of docetaxel, oxaliplatin and S1 (DOS) to patients with gastric cancer.

DETAILED DESCRIPTION:
The primary aim of this dose-finding study is to determine the maximum tolerated doses of docetaxel, oxaliplatin and S1 given every second (DOS2w) or third (DOS3w) week as first-line treatment in patients with advanced gastro-esophageal cancer. Secondary end points are to evaluate toxicities according to NCI-CTCAE v. 4, response rate, progression-free survival and overall survival

Primary Outcome Measure:

To determine maximum tolerated dose (MTD) for the the combination regimes (DOS2w) and (DOS3w).

The investigators have planned to examine 4 dose levels of (DOS2w) and 3 dose levels of (DOS3w).

Methods:

This dose-finding study is planned to include a total of 24 patients with advanced gastro-esophageal cancer, adenocarcinoma.

12 patients will be included in (DOS2w) at four at progressively higher dose levels.

Chemotherapy will be repeated day 1 every second week to a maximum of nine courses.

12 patients will be included in (DOS3w) at three progressively higher dose levels.

Chemotherapy will be repeated day 1 every third week to a maximum of six courses.

In both (DOS2w) and (DOS3w) dose-limiting toxicity (DLT) will be evaluated after the first course. In case of DLT among one of the three patients during the first course of treatment additional three patients will be added at the respective dose level. Dose escalation is continues if 0/3 or 1/6 patients experience DLT.

Patients will be evaluated with a ct-scan at baseline and after every three or four cycles to exclude progression and evaluate response. Response is assessed by the investigator according to RECIST version 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven adenocarcinoma of the esophagus or the ventricle (ECV), and which cannot be treated curatively.
2. Age ≥ 18 years.
3. WHO performance status 0-1.
4. Neutrophils ≥ 1,5 x 109/L and platelets ≥ 100 x 109/L.
5. Bilirubin ≤ 1,5 x UNL (Upper Normal Limit) and ASAT and/or ALAT ≤ 3 x UNL.
6. Creatinine-clearance ≥ 60 ml/min.
7. Planned first day of treatment within 8 days after inclusion in the study.
8. Signed consent form.

Exclusion Criteria:

1. No previous treatment with chemotherapy, except for (neo)-adjuvant chemotherapy for adenocarcinoma - treatment should have been completed at least 6 months before entrance in this study.
2. No sensory neuropathy.
3. No previously treatment with docetaxel, oxaliplatin or S1.
4. No clinical suspicion of brain metastases.
5. No cytotoxic treatment or other experimental treatment within 2 weeks of inclusion in the study.
6. Other serious disease (i.e. heart disease, AMI within 1 year or ongoing infection).
7. No pregnant women or women who are lactating. Patients who are not using contraception.
8. No known DPD-deficiency or known allergy to taxanes or platinum.
9. No signs of physical or mental illness that would prevent absorption of oral treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06-05 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, Professor, Study Chair — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Result] Pfeiffer P, Qvortrup C, Krogh M, Schoennemann K, Vestermark LW, Jensen HA, Bjerregaard JK. S-1 in combination with docetaxel and oxaliplatin in patients with advanced gastro-esophageal adenocarcinoma: two parallel phase 1/2a studies. Acta Oncol. 2017 Jan;56(1):46-51. doi: 10.1080/0284186X.2016.1257865. Epub 2016 Dec 2. PMID 27911128

RESULTS

PARTICIPANT FLOW:
Groups:
- DOS2w 1A: 3 patients Docetaxel mg/m2 day 1: 30 Oxaliplatin mg/m2 day 1: 70 S-1 mg/m2 days 1-7: 30x2
- DOS2w 2A: 3 patients Docetaxel mg/m2 day 1: 30 Oxaliplatin mg/m2 day 1: 70 S-1 mg/m2 days 1-7: 35x2
- DOS 2w 3A: 6 patients Docetaxel mg/m2 day 1: 40 Oxaliplatin mg/m2 day 1: 70 S-1 mg/m2 days 1-7: 35x2
- DOS2w 4A: 6 patients Docetaxel mg/m2 day 1: 50 Oxaliplatin mg/m2 day 1: 70 S-1 mg/m2 days 1-7: 35x2
- DOS3w 1B: 3 patients Docetaxel mg/m2 day 1: 40 Oxaliplatin mg/m2 day 1: 100 S-1 mg/m2 days 1-7: 25x2
- DOS3w 2B: 8 patients Docetaxel mg/m2 day 1: 50 Oxaliplatin mg/m2 day 1: 100 S-1 mg/m2 days 1-7: 25x2
- DOS3w 3B: 5 patients Docetaxel mg/m2 day 1: 60 Oxaliplatin mg/m2 day 1: 100 S-1 mg/m2 days 1-7: 25x2
Period: Overall Study
Arm/Group | DOS2w 1A | DOS2w 2A | DOS 2w 3A | DOS2w 4A | DOS3w 1B | DOS3w 2B | DOS3w 3B
Started | 3 | 3 | 6 | 6 | 3 | 8 | 5
Completed | 3 | 3 | 6 | 6 | 3 | 8 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DOS2W Dose Level 1A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (60 mg/m2) will be given every 2nd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS3W Dose Level 1B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (40 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS2W Dose Level 2A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS2W Dose Level 3A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (40 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS2W Dose Level 4A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (50 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS3W Dose Level 2B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (50 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- DOS3W Dose Level 3B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (60 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week. In total there is 5 dose levels and if no patients experience DLT on a given level, next dose level will be administered.
- Total: Total of all reporting groups
Arm/Group | DOS2W Dose Level 1A | DOS3W Dose Level 1B | DOS2W Dose Level 2A | DOS2W Dose Level 3A | DOS2W Dose Level 4A | DOS3W Dose Level 2B | DOS3W Dose Level 3B | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 8 | 5 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 2 | 4 | 2 | 3 | 3 | 17
  >=65 years | 1 | 2 | 1 | 2 | 4 | 5 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 5 | 3 | 1 | 3 | 12
  Male | 3 | 3 | 3 | 1 | 3 | 7 | 2 | 22
Region of Enrollment [Number; unit: participants]
  Denmark | 3 | 3 | 3 | 6 | 6 | 8 | 5 | 34

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival
Time Frame: Up to 2 years after first administration of DOS
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- DOS2W 1A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (60 mg/m2) will be given every 2nd week.
- DOS2W 2A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
- DOS2W 3A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (40 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
- DOS2W 4A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2W: Docetaxel (50 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
- DOS3W 1B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (40 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week.
- DOS3W 2B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (50 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week.
- DOS3W 3B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3W: Docetaxel (60 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 3rd week.
Arm/Group | DOS2W 1A | DOS2W 2A | DOS2W 3A | DOS2W 4A | DOS3W 1B | DOS3W 2B | DOS3W 3B
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 3 | 8 | 5
Months | 4.3 [1 to 8] | 13.8 [7 to 16] | 14.6 [7 to 25] | 15.2 [6 to 26] | 8.3 [5 to 12] | 16.4 [8 to 24] | 7.8 [4 to 13]

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- DOS2w Dose Level 1A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2w: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (60 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS2w Dose Level 2A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2w: Docetaxel (30 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS2w Dose Level 3A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2w: Docetaxel (40 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS2w Dose Level 4A: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS2w: Docetaxel (50 mg/m2), Oxaliplatin (70 mg/m2) and S1 (70 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS3w Dose Level 1B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 3rd week.
  DOS3w: Docetaxel (40 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS3w Dose Level 2B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS3w: Docetaxel (50 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
- DOS3w Dose Level 3B: Treatment with Docetaxel, Oxaliplatin and S1. Treatment is given every 2nd week.
  DOS3w: Docetaxel (60 mg/m2), Oxaliplatin (100 mg/m2) and S1 (50 mg/2) will be given every 2nd week.
  Dose levels are described in the Participant Flow section.
Arm/Group | DOS2w Dose Level 1A | DOS2w Dose Level 2A | DOS2w Dose Level 3A | DOS2w Dose Level 4A | DOS3w Dose Level 1B | DOS3w Dose Level 2B | DOS3w Dose Level 3B
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 3/6 | 3/6 | 3/3 | 6/8 | 4/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/6 | 2/6 | 0/3 | 1/8 | 2/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 4/6 | 0/6 | 0/3 | 1/8 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOS2w Dose Level 1A (N=3) | DOS2w Dose Level 2A (N=3) | DOS2w Dose Level 3A (N=6) | DOS2w Dose Level 4A (N=6) | DOS3w Dose Level 1B (N=3) | DOS3w Dose Level 2B (N=8) | DOS3w Dose Level 3B (N=5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOS2w Dose Level 1A (N=3) | DOS2w Dose Level 2A (N=3) | DOS2w Dose Level 3A (N=6) | DOS2w Dose Level 4A (N=6) | DOS3w Dose Level 1B (N=3) | DOS3w Dose Level 2B (N=8) | DOS3w Dose Level 3B (N=5)
Diarrhea grade 3-4 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea grade 3-4 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting grade 3-4 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue grade 3-4 (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy grade 3-4 (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No